CLINICAL TRIAL: NCT06406062
Title: To Evaluate the Effectiveness and Safety of an Artificial Intelligence-assisted System in Colonoscopy in a Real-world Obsevational Multicenter Study
Brief Title: Artificial Intelligence-assisted System in Colonoscopy
Status: Recruiting | Type: Observational
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024K-K017
Record Dates: First submitted 2024-04-25; First posted 2024-05-09 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Adenoma Colon Polyp

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- AI-assisted group: Group with AI assistance
  Interventions: Device: ANDOANGEL
- Control group: Group without AI assistance

INTERVENTIONS:
Device: ANDOANGEL — Polyps were identified by endoscopists assisted by an AI system: rectangular box marks; Monitoring of ileocecal position: whether blindness was reached was displayed in the lower left corner of the interface.
  Mirror entry and exit time monitoring: the operation time is displayed in the upper left corner of the interface.
  Colonoscopy withdrawal speed monitoring: the relative withdrawal speed was displayed on the left side of the interface.
  Groups: AI-assisted group

SUMMARY:
In recent years, computer-aided diagnosis system based on artificial intelligence (AI) has been used in colorectal polyp detection. In recent years, computer-aided diagnosis system based on artificial intelligence (AI) has been used in colorectal polyp detection. However, whether AI-assisted can improve the adenoma-detection rate (ADR) is inconclusive. This study aims to evaluate the real-world performance of an AI system that combines polyp detection with colonoscopy quality control.

This study aims to explore the clinical application value of AI-based polyp detection and quality control function by comparing the data of polyp detection rate and adenoma detection rate in multiple centers with and without AI-assisted colonoscopy in a multicenter, prospective real world study. However, whether AI-assisted can improve the adenoma-detection rate (ADR) is inconclusive. This study aims to evaluate the real-world performance of an AI system that combines polyp detection with colonoscopy quality control.

This study aims to explore the clinical application value of AI-based polyp detection and quality control function by comparing the data of polyp detection rate and adenoma detection rate in multiple centers with and without AI-assisted colonoscopy in a multicenter, prospective real world study.

ELIGIBILITY:
Inclusion Criteria:

1. age > 50 years old;
2. required diagnostic colonoscopy, screening colonoscopy, or follow-up colonoscopy;
3. voluntarily sign informed consent;
4. Commitment to abide by the study procedures and cooperate with the implementation of the whole process of the study.

Exclusion Criteria:

1. have participated in other clinical trials, signed informed consent and are in the follow-up period of other clinical trials;
2. known polyposis syndrome patients;
3. patients with known IBD;
4. patients considered by the investigators to be unsuitable or unable to undergo complete digestive endoscopy and related examinations;
5. high-risk diseases or other special conditions considered by the investigator to be unsuitable for clinical trial participation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients required diagnostic colonoscopy, screening colonoscopy, or follow-up colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | During Endoscopy procesure
  The numerator is the number of patients who had at least one adenoma on colonoscopy, and the denominator is the total number of patients who underwent colonoscopy

SECONDARY OUTCOMES:
Polyp detection rate | During Endoscopy procesure
  The numerator is the number of patients who had at least one polyp on colonoscopy, and the denominator is the total number of patients who underwent colonoscopy
Detection rate of serrated adenoma | During Endoscopy procesure
  The numerator is the number of patients who had at least one serrated adenoma on colonoscopy, and the denominator is the total number of patients who underwent colonoscopy
Average number of polyps per colonoscopy | During Endoscopy procesure
  The numerator is the total number of polyps detected by colonoscopy, and the denominator is the total number of colonoscopies
Colonoscopy time | During Endoscopy procesure
  The pure negative time of the whole examination did not include the time of endoscopy entry and the time of biopsy
Proportion of over-speed frames | During Endoscopy procesure

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan Univercity, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No